CLINICAL TRIAL: NCT04403438
Title: Pain, Sleep, Fatigue, Physical Activity Level, Quality of Life and Exercise Habits in Patients With Familial Mediterranean Fever and Behçet: Analysis Before and After Covid19 Pandemic
Brief Title: Familial Mediterranean Fever and Behçet: Analysis Before and After Covid19 Pandemic
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nejla Uzun, MSc, Pt, Istanbul University
Other Study IDs: 10840098-604.01.01-E.14697
Record Dates: First submitted 2020-05-23; First posted 2020-05-27 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2023-06

CONDITIONS: Behcet Disease; COVID; FMF
MeSH Terms: conditions — Behcet Syndrome | interventions — Sleep; Quality of Life; Pyrin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with behçet's or fmf
  Interventions: Other: ıt will be compared pain, sleep, fatigue, physical activity level and quality of life and questioning exercise habits before and after the covid-19 outbreak in patients with Behçet and FMF.

INTERVENTIONS:
Other: ıt will be compared pain, sleep, fatigue, physical activity level and quality of life and questioning exercise habits before and after the covid-19 outbreak in patients with Behçet and FMF. — ıt will be compared pain, sleep, fatigue, physical activity level and quality of life and questioning exercise habits before and after the covid-19 outbreak in patients with Behçet and FMF.

SUMMARY:
Behcet' disease (BD) is a chronic inflammatory disease which is characterized by oral and genital ulcers, uveitis and skin lesions. Musculoskeletal involvement such as arthrits, arthralgia, enthesis and sacroiliitis can be seen in course of BD. FMF is an autosomal recessive family disease characterized by abdominal pain, chest pain, joint pain and fever attacks as a result of inflammation of the serous membranes. FMF patients have been shown to experience higher levels of pain, fatigue, depression and anxiety than healthy controls, and this has increased sleep disturbance and reduced quality of life. FMF and BiH have common characteristics such as ethnicity, etiopathogenetic mechanisms, symptoms, and treatment. In December 2019, after the officially detected coronavirus (severe acute respiratory syndrome coranavirus-2 [SARS-CoV-2]) resistant to unknown treatment and rapidly spreading coronavirus in our country on March 11, 2020 in Hubei province of China, the number of cases increased rapidly and virus was isolated in 670 patients within 10 days. Ongoing concerns about the spread of Covid-19 infections have caused many measures to be taken. Among them, social isolation, home quarantine and avoiding collective places are the most important. In our country, in the process of social isolation, the areas of movement of Behçet and FMF patients, like everyone else, were restricted, their stress and anxiety levels increased and their motivation decreased. The aim of our study is to compare the pain, sleep, fatigue, physical activity level and quality of life and question exercise habits before and after the covid-19 outbreak in patients with Behçet and FMF.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Being diagnosed with FMF at least 1 year ago according to diagnostic criteria
* A diagnosis of BiH at least 1 year ago according to the International Behçet Working Group
* Having signed the informed consent form
* Having a cooperative level that will respond to evaluation scales

Exclusion Criteria:

* Pregnant women
* Having other chronic diseases
* Psychiatric disorders and treated
* Those with cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In patients with Behçet and FMF between the ages of 18-65, exercise habits will be questioned by comparing pain, sleep, fatigue, physical activity level and quality of life before and after the covid-19 outbreak.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
IPAQ-SF | one assesment baseline
  The Turkish validity and reliability study of this short questionnaire consisting of seven questions, which evaluates in detail the amount of walking performed in the last week and the amount of moderate and difficult physical activity performed in work, transportation, housework, gardening and leisure activities.
Numeric Rating Scale | one assesment baseline
  It has horizontal and vertical forms. In this scale, the starting point is the point where there is no pain, and the ending point is the end point where the pain is worst

SECONDARY OUTCOMES:
Short-Form 36 Health Survey (SF-36) | one assesment baseline
  It is a scale which was found by Ware in 1987 and examined the quality of life of people. Turkish validity was provided in the study of Koçyiğit et al. The scale consisting of 36 questions was divided into its own subtitles and was made to measure the functional status of the person.
Exercise Stage of Change Questionnaire | one assesment baseline
  it consists of five questions. The participant is asked to choose only one of these five situations that match the current exercise level.
Exercise Self-Efficacy Questionnaire | one assesment baseline
  This six-point five-point Likert-type scale determines the self-confidence of individuals to begin exercise. The lowest 6 and the highest 30 points are obtained from the scale. The high scores obtained from the scale indicate that the individual trusts him / herself and has a high chance of success in change.
Decisional Balance Questionnaire | one assesment baseline
  Items 2, 4, 6, 8, 10 on a scale consisting of a total of 10 items are expressions designed to evaluate the perceived harm of not exercising, items 1, 3, 5, 7, and 9 are intended to evaluate the perceived benefits of exercising.

CONTACTS AND LOCATIONS:
Overall Officials: nejla uzun, MSc, Pt, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- IstanbulU, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No